CLINICAL TRIAL: NCT04605432
Title: Face-to-face Instructions and Personalized Bowel Cleansing Regimens for Inpatients Could Improve Bowel Preparation Quality.
Brief Title: FFI and PR Could Improve Bowel Cleansing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FFI-1.0
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-01

CONDITIONS: Bowel Preparation
Keywords: bowel preparation; face-to-face instruction; personalized intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-FFI prep (Experimental): On the day before colonoscopy, an experienced researcher would go to the ward to have a face-to-face conversation with the patient to know if patients have the risk factors for bowel preparation failure.
  The bowel preparation regimens for patients with risk factors would be optimized. In addition to drink single dose of 120g Polyethylene Glycol (PEG-4000) with 3L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min, the patient also drink single dose of 60g Polyethylene Glycol (PEG-4000) with 1L water at 20:00- 21:00 hours on the day before the colonoscopy. Patients without risk factors drink single dose of 120g Polyethylene Glycol (PEG-4000) with 3L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Patients would received a booklet to explain the details of diet restriction, preparation method and the pictures of bowel preparation of results.The researcher would give a detailed oral explanation of the booklet.
  Interventions: Drug: PEG-FFI
- PEG-nonFFI prep (Active Comparator): Patients in the PEG-nonFFI group would only receive routine patient education on bowel preparation of colonoscopy, which was completed by ward nurse. all the patients drink single dose of 120g Polyethylene Glycol (PEG-4000) with 3L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Interventions: Drug: PEG-nonFFI

INTERVENTIONS:
Drug: PEG-FFI — Patients with risk factor : on the day before the colonoscopy at 20:00- 21:00 hours, 60gPEG-4000 was mixed with 1L water; 4-6 h before colonoscopy, 120gPEG-4000 was mixed with 2L water.
  Patient without risk factor: 4-6 hours before colonoscopy, 120gPEG-4000 was mixed with 3L water.
  Education completed by experienced researcher.
  Arms: PEG-FFI prep
Drug: PEG-nonFFI — All patients on the day of the colonoscopy:4-6 hours before colonoscopy, 120gPEG-4000 was mixed with 3L water.
  Education completed by ward nurse.
  Arms: PEG-nonFFI prep

SUMMARY:
background:The use of enhanced instruction can improve the efficiency of education for bowel preparation regimens. Researchers hypothesized that face-to-face instruction and personalized intervention for inpatient could improve successful bowel preparation rate and patient's compliance with regimens.

Methods:This was an endoscopist-blind,randomized controlled trial. 320inpatients were randomized 1:1 in one of the two study groups. The intervention group received face-to-face instruction and personalized intervention for bowel preparation protocol, while control group received the standard bowel preparation protocol. Patients'demographics, bowel preparation quality, colonoscopy completion and attendance were recorded. Logistic regression was performed to identify predictors of bowel preparation failure.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients undergoing colonoscopy.
* patients older than 18 years.

Exclusion Criteria:

* prior surgery of colorectal resection;
* suspected colonic stricture or perforation;
* incomplete or complete bowel obstruction;
* use of prokinetic agents or purgatives within 7 days;
* Patients with severe gastrointestinal diseases, such as intestinal obstruction or perforation, active ulcerative colitis, toxic colitis and toxic megacolon;;
* pregnancy or lactation;
* Inability to prepare bowel;
* unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | 1 Day of colonoscopy
  The BBPS is a validated scoring system with scores between 0 and 9, where 9 is the best score. The score comprises a sub score 0-3 for each colon segment: right, transverse and left colon.
  For all participants, BBPS score will be used when colonscopy is withdrawing.

SECONDARY OUTCOMES:
adverse events | The day of colonoscopy and the day before
  Including nausea, vomiting, abdominal pain and bloating,etc.
cecal intubation rate | 1 Day of colonoscopy
  The number of colonoscopy reaching the cecal area divided by the total number of colonoscopy
polyp detection rate | 1 Day of colonoscopy
  PDR was defined as the number of patients with at least one polyp divided by the total number of colonoscopy patients
cecal intubation time | 1 Day of colonoscopy
  Time to reach the cecal
withdrawal time | 1 Day of colonoscopy
  Time from withdrawal from the cecum to the end of colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo No. 1 Hospital, Ningbo, Zhejiang, China